CLINICAL TRIAL: NCT00001147
Title: Blood Sampling for Neurochemical and Genetic Testing
Status: Completed | Type: Observational
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000008; 00-N-0008
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2004-03

CONDITIONS: Autonomic Nervous System Disease; Healthy; Hypertension; Pheochromocytoma
Keywords: Dopamine; Metanephrine; Norepinephrine; Epinephrine; Catecholamines; Tyrosine Hydroxylase; Monoamine Oxidase; Phenosulfotransferase; Sympathetic Nervous System; Normetanephrine
MeSH Terms: conditions — Hypertension; Pheochromocytoma

SUMMARY:
This study involves sampling blood from both normal volunteers and patients with diseases known or suspected to involve body chemicals called catecholamines. The blood will be used to establish normal values for plasma levels of catecholamines and related neurochemicals; to test for abnormal neurochemical patterns in patients; and to establish a "bank" of DNA from normal volunteers and from patients to be used in future studies about possible alterations of catecholamine-related genes.

Study participants will report to NIH after fasting overnight except for water or noncaloric, noncaffeinated beverages. They must not have taken Tylenol for at least 5 days. Blood will then be drawn. DNA will be extracted and stored in the freezer for future studies.

DETAILED DESCRIPTION:
This project is to allow blood sampling from normal volunteers and patients with dysautonomia, pheochromocytoma, hypertension, or neurogenetic diseases involving catecholaminergic systems. The blood is used to establish normal values for plasma levels of catechols and related neurochemicals; test for abnormal neurochemical patterns in patients; and establish a "bank" of DNA samples from normal volunteers and from patients, to be used in future studies about mutations or polymorphisms of catecholamine-related genes.

ELIGIBILITY:
INCLUSION CRITERIA:

The subjects are healthy normal volunteers or patients with dysautonomia, pheochromocytoma, hypertension, or neurogenetic diseases involving catecholaminergic systems. Children of any age above 4 years may participate. In the case of minors, consent is obtained from an adult who is legally responsible for the subject.

EXCLUSION CRITERIA:

Subjects in whom anatomic or technical factors preclude insertion of an arm intravenous (i.v.) catheter are excluded. Normal volunteers taking any prescribed medication are excluded. Normal volunteers who smoke cigarettes or consume alcohol daily are excluded.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 500
Dates: Start 1999-10; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Neurological Disorders and Stroke (NINDS), Bethesda, Maryland, United States

REFERENCES:
- [Background] Goldstein DS, Lenders JW, Kaler SG, Eisenhofer G. Catecholamine phenotyping: clues to the diagnosis, treatment, and pathophysiology of neurogenetic disorders. J Neurochem. 1996 Nov;67(5):1781-90. doi: 10.1046/j.1471-4159.1996.67051781.x. PMID 8863481